CLINICAL TRIAL: NCT03024008
Title: A Multicenter Study to Evaluate the Enhancement of Bone Regeneration and Healing in the Extremities by the Use of Autologous BonoFill-II
Brief Title: Enhancement of Bone Regeneration and Healing in the Extremities by the Use of Autologous BonoFill-II
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BonusBio Group Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-BNS05
Record Dates: First submitted 2017-01-11; First posted 2017-01-18 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-08

CONDITIONS: Bone Fracture
Keywords: Critical Gap; Comminuted Fracture; Extra-Articular
MeSH Terms: conditions — Fractures, Bone; Fractures, Comminuted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Clinical Interventions:
  1. Blood tests: complete blood count, full blood chemistry and biochemistry including phosphate, alkaline phosphatase, calcium, renal and liver function, and coagulation. Serology tests: HIV, Hepatitis B, Hepatitis C.
  2. Xray
  3. Urine Test
  4. CT
  5. Liposuction - harvest of 50-300ml autologous adipose tissue from the subject's abdomen
  6. Single transplantation of Investigational Medicinal Product BonoFill-II into long bone extra-articular comminuted fracture or large bone defect/critical gap
  Interventions: Biological: BonoFill-II

INTERVENTIONS:
Biological: BonoFill-II — Surgery will be performed under local or general anesthetics according to the Investigator's and anesthesiologist discretion.
  A standard orthopedic approach will be made according to the fracture site.Then the transplantation of BonoFill-II into the fracture site and the fixation of the fracture by intramedullary nail or plate and screws or external fixator as required will be performed.
  internal fixation (plate and screws and intramedullary nails) will not be routinely removed. External fixators will be removed upon achievement of satisfactory bone union.

SUMMARY:
The purpose of this clinical study is to evaluate the safety and the efficacy of BonoFill-II as an autologous bone-regenerating graft in the reconstruction of deficient bone in two clinical indications:

1. Long and short bone extra-articular comminuted fracture
2. Long and short bones extra and intra articular defect /Gap or non-union, incapable of self-regeneration

DETAILED DESCRIPTION:
Primary Endpoint:

Safety: to establish that the transplantation of BonoFill-II into bone defect/gap is safe under the following conditions:

* No treatment-related appearance of heterotrophic bone ossification
* No excessive bone formation at the transplantation sites
* No abnormalities in the treated sites

Efficacy: to establish that the transplantation of BonoFill-II into bone defect/gap is effective under the following conditions:

* Bone continuity, measured radiographically by CT at 6 and 12 months.
* Weight-bearing ability, assessed at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Long and short bones extra articular comminuted fracture or
* Long and short bones extra and intra articular defect/gap or non union, incapable of self-regeneration

Exclusion Criteria:

* Age is under 18 or above 80
* A simple fracture manageable by one definitive treatment
* Pregnant or lactating women
* Patients with active infection that is in question and needs osteogenic treatment.
* More than 3 previous failed interventions at the surgical site
* History of advanced congestive heart failure or active acute myocardial infarction (AMI), renal failure (estimated GFR of <30 ml/min/1.73 m2 at screening), or hepatic disease (hepatic insufficiency classified as Child-Pugh B or C)
* Diabetic subjects (HbA1c > 8)
* Subject treated currently with systemic steroids.
* Subjects with known autoimmune diseases, such as Addison's disease, Celiac disease - sprue (gluten-sensitive enteropathy), Dermatomyositis, Graves disease, Hashimoto's thyroiditis, Multiple sclerosis, Myasthenia gravis, Pernicious anemia, Reactive arthritis, Rheumatoid arthritis, Sjogren syndrome, Systemic lupus erythematosus.
* Subjects diagnosed with osteoporosis
* Chronic severe PVD (Peripheral Vascular Disease) subjects
* Post major vascular operation in the treated limb/s and above the surgical site (with or without Gore-Tex grafting)
* Subjects that have a known scar healing problem (keloid formation).
* Subjects treated with Bisphosphonate drugs
* Oncology patient or subjects who received chemotherapy or radiotherapy treatment in the past 12 months
* Immunocompromised condition from any reason, at screening
* Subjects participating in another clinical trial 30 days prior to and during the study period.
* Drug addicts and psychiatric patients patients incapable of giving consent.
* Subjects with a known history of any significant medical disorder, which in the investigator's judgment contraindicates the subject's participation
* Subjects with any known allergy for local/general anesthesia
* Positive serology for either HIV, hepatitis B or hepatitis C
* Abnormal clinically significant laboratory test and findings, as per the investigator's judgment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint: Absence of treatment-emergent appearance of safety issues | Throughout the post-intervention 12-month follow-up
  Subjects demonstrating no appearance of heterotrophic bone ossification, excessive bone formation and/or any abnormalities in the treated site, in the proximal or distal joint by visual examination of the transplantation site and by X-ray and/or CT.
Efficacy endpoint: Bone continuity | Starting 4-week follow-up and through to the end of the 12-month follow-up
  Bone union, as assessed by X-ray and CT. CT scans are performed 6 and 12 months post operation, to verify bone regeneration and complete bone continuity was achieved.
Functional efficacy endpoint: Weight bearing ability | The test is performed at 3, 6 and 12 months post operation.
  clinical examination of weight bearing ability for lower extremities or coffee-cup weight bearing ability for upper extremities. The physician assesses the functionality of the operated limb, by testing the patients ability to bear their weight when standing (in case of lower limb bone defect) or by coffee cup holding simulation (in case of upper limb bone defect).

OTHER OUTCOMES:
Lack of pain at the surgical site | 3, 6 and 12 months
  Pain at the surgical site will be evaluated using a VAS pain scale, this assessment will be used in cases of bone defect where weight-bearing is not applicable due to further limb injuries (such as nerve injuries or other non-bone defects).

CONTACTS AND LOCATIONS:
Overall Officials: Nimrod Rozen, MD, PhD, Principal Investigator — Emek Medical Center, Afula, Israel
Locations (6):
- Israel (6):
  - Emek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Hillel Yafe, Hadera
  - Carmel Medical Center, Haifa
  - Rambam Health Campus, Haifa
  - Meir Medical Center, Kfar Saba

IPD SHARING:
Plan to Share IPD: No